CLINICAL TRIAL: NCT02570594
Title: Autobiographical Memory Organization in Schizophrenia
Acronym: AMOrSchiz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5506
Record Dates: First submitted 2013-02-12; First posted 2015-10-07 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Cognition; Autobiographical; memoryCognitive; remediation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Other)
  Interventions: Other: questionary

INTERVENTIONS:
Other: questionary

SUMMARY:
The aim of the study is to investigate the temporal organization of autobiographical memory in patients with schizophrenia. Patients and control participants will be invited separately to participate in a 1hour walk in the city of Strasbourg and at the same time, to carry an automatic camera around their neck, which is called SenseCam®. Pictures obtained with SenseCam® will be later presented to the participants during the session of test. They will be asked to determine the chronological order of 12 pictures corresponding to 12 particular events of the tour. Then they will be asked to watch the complete sequence of photos from the tour and to determine the beginning and ending of the events that have occurred during the tour. According to the investigators hypotheses, patients should have difficulty to find out the correct chronological order of the photos and to determine the appropriate beginnings and endings of the events

ELIGIBILITY:
Inclusion Criteria:

* for both patients and controls
* male or female willing to participate and who have signed up the legal document
* under the protection of health insurance for patients only
* schizophrenia or schizo-affective disorder according to the DSM-IV-TR criteria
* clinically stable for at least 2 months for controls only
* no psychiatric history

Exclusion criteria:

* for both patients and controls
* current severe or unstable somatic illness
* neurological history (epilepsia, brain injury, brain surgery…)
* current substance use disorder (DSM-IV-TR)
* current major depressive disorder (DSM-IV-TR)
* mental retardation (IQ < 70)
* pregnancy, breast feeding
* current legal control for patients only
* treatment comprising benzodiazepines
* benzodiazepines intake during the last 3 weeks for controls only
* psychotropic intake during the last 3 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Specificity of memories recovered by using the SenseCam camera during the trial | 1 month
  SenseCam®(corresponding to the name of the automatic camera that participants will be asked to carry around their neck during the city-tour)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de psychiatrie 1 , Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France

REFERENCES:
- [Result] Alle MC, Giersch A, Potheegadoo J, Meyer N, Danion JM, Berna F. From a Lived Event to Its Autobiographical Memory: An Ecological Study Using Wearable Camera in Schizophrenia. Front Psychiatry. 2019 Oct 4;10:699. doi: 10.3389/fpsyt.2019.00699. eCollection 2019. PMID 31636574